CLINICAL TRIAL: NCT00751816
Title: Head & Neck Cancer Survivorship: Physical and Functional Status
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000613863; VU-VICC-SUPP-0843
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Head and Neck Cancer
Keywords: musculoskeletal complications; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; stage I adenoid cystic carcinoma of the oral cavity; stage I mucoepidermoid carcinoma of the oral cavity; stage I verrucous carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage I basal cell carcinoma of the lip; stage II basal cell carcinoma of the lip; stage III basal cell carcinoma of the lip; stage IV basal cell carcinoma of the lip; stage I lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; high-grade salivary gland mucoepidermoid carcinoma; low-grade salivary gland mucoepidermoid carcinoma; salivary gland acinic cell tumor; salivary gland adenocarcinoma; salivary gland adenoid cystic carcinoma; salivary gland anaplastic carcinoma; salivary gland malignant mixed cell type tumor; salivary gland poorly differentiated carcinoma; salivary gland squamous cell carcinoma; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms | interventions — Neoadjuvant Therapy; Chemotherapy, Adjuvant; Physical Therapy Modalities; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Supportive Care: head and neck cancer survivors who are undergoing chemotherapy and radiation therapy
  Interventions: Drug: systemic chemotherapy; Other: survey administration; Procedure: adjuvant therapy; Procedure: management of therapy complications; Procedure: musculoskeletal complications management/prevention; Procedure: physical therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: systemic chemotherapy
  Other Names: none noted
Other: survey administration — will be administered before, during, and after medical intent-to-cure treatment to describe head and neck cancer survivors' physical and functional well-being.
  Other Names: none noted
Procedure: adjuvant therapy
  Other Names: none noted
Procedure: management of therapy complications
  Other Names: None noted
Procedure: musculoskeletal complications management/prevention
  Other Names: none noted
Procedure: physical therapy — weekly visits coordinated with adjuvant treatment as part of standard care
  Other Names: none noted
Radiation: radiation therapy
  Other Names: none noted

SUMMARY:
RATIONALE: Early physical therapy may be effective in improving range of motion of the neck and shoulders in head and neck cancer survivors who are undergoing chemotherapy and radiation therapy.

PURPOSE: This phase I trial is studying how well early physical therapy works in improving physical and functional well-being in head and neck cancer survivors receiving chemoradiotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Describe the physical and functional well-being of head and neck cancer (HNC) survivors undergoing physical therapy during adjuvant chemoradiotherapy.
* Describe clinical measure of range of motion for the cervical spine and shoulder of HNC survivors undergoing physical therapy during adjuvant chemoradiotherapy.
* Determine the feasibility of an early physical therapy intervention (prior to and during adjuvant treatment) targeting the physical needs of HNC survivors.

OUTLINE: Patients undergo physical therapy weekly for 10 weeks beginning 1 week prior to initiating adjuvant chemoradiotherapy and continuing until 2 weeks after the completion of adjuvant chemoradiotherapy.

Patients undergo range of motion assessment and complete a Cancer Survivorship Survey (CSS) at baseline and in weeks 4, 8, 9, and 10 of physical therapy.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Head and neck cancer survivor
* Planning to receive adjuvant chemoradiotherapy for head and neck cancer

  * Has not yet initiated adjuvant therapy
* Referred to rehabilitation oncology physical therapy program

Exclusion Criteria:

* No metastatic disease
* No CNS cancer

PATIENT CHARACTERISTICS:

* Speaks English
* No significant history of cardiovascular or neurovascular disease involving disability

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Not currently in hospice care

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head and Neck Cancer Patients
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2008-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Physical and functional well-being during adjuvant chemoradiotherapy | 2 weeks after completing treatment
Range of motion for the cervical spine and shoulder during adjuvant chemoradiotherapy | 2 weeks after completing treatment
Feasibility of an early physical therapy intervention | 2 weeks after completing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ann Marie Flores, Ph.D., Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee